CLINICAL TRIAL: NCT00921128
Title: Convection Enhanced Delivery of Muscimol to Study the Pathophysiology Underlying the Clinical Features of Parkinson's Disease
Brief Title: Convection-Enhanced Delivery to Study the Pathophysiology Underlying the Clinical Features of Parkinson s Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090160; 09-N-0160
Record Dates: First submitted 2009-06-13; First posted 2009-06-16 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2016-09-01

CONDITIONS: Parkinson's Disease
Keywords: Muscimol; Convection-Enhanced Delivery; Parkinson's Disease; Deep Brain Stimulation; Parkinson Disease; PD
MeSH Terms: conditions — Parkinson Disease | interventions — Muscimol

INTERVENTIONS:
Drug: Muscimol

SUMMARY:
Background:

* Parkinson s disease (PD) is a progressive neurodegenerative disorder that affects the brain cells that make the chemical dopamine. The primary medical treatment for PD has been to use medications to replace the dopamine that is missing from the brain. These medications can be effective at first, but after many years side effects and tolerance develop.
* Surgery can treat basic PD symptoms and complications. Deep brain stimulation (DBS) offers a safer alternative as the therapy can be adjusted and reversed to minimize side effects and optimize beneficial effects. DBS treats the symptoms of PD but does not alter its course.
* Infusions of neurochemicals or medications are another PD treatment method. NIH researchers have developed the technique of convection-enhanced delivery, which very precisely and consistently delivers infusions of many types into the brain. This project will allow researchers to infuse a medication, Muscimol, into the subthalamic region of the brain to see if it is as safe and effective as DBS.

Objectives:

* To determine whether an infusion of Muscimol into the brain is safe and relieves the symptoms of Parkinson s disease.
* To demonstrate that the infusion can be monitored with magnetic resonance imaging (MRI) using gadolinium.

Eligibility:

* Patients 18 years of age and older who have Parkinson s disease and are preparing for bilateral subthalamic nucleus (STN) DBS surgery.
* Patients will be divided into two groups. One group of patients will have a partial infusion of Muscimol into the STN, and the second group of patients will have complete infusion of Muscimol into the STN.

Design:

* This study will begin 5 days before the patient undergoes bilateral subthalamic DBS surgery.
* On Day 1 of the study, small thin tubes (microcatheters) will be inserted into the STN through the same incision and burr holes that are used for DBS. Two infusion studies of Muscimol will be performed on successive days: the first without PD medication (Day 3 of study) and the second with PD medication (Day 4 of study).
* Each infusion will be monitored in the MRI suite, and researchers will perform clinical examinations of patients PD symptoms.
* Following the study experiments, a second surgery will be performed to remove the microcatheters and to place DBS electrodes in the standard fashion.

DETAILED DESCRIPTION:
Objective: The objectives of this pilot study are to gain insight into the safety, feasibility and clinical effects of infusion of a temporary acting GABAA agonist (muscimol) by convection-enhanced delivery into the subthalamic nuclei (STN) of Parkinson s disease (PD) patients undergoing deep brain stimulation (DBS) surgery.

Study population: Eight adult male and female patients with medically-intractable PD who are preparing to undergo DBS surgery and who meet all Inclusion and Exclusion Criteria will be enrolled. Six subjects will be treated (2 may be screening failures).

Design: We propose a single center pilot study of infusion of muscimol into the bilateral STN of PD patients that will undergo DBS. Subjects will be enrolled into 1 of 2 cohorts. Both cohorts will contain 3 patients each (total of 6 patients). Patients in both cohorts will undergo pre-, intra- and post-operative PD assessments. The first cohort will undergo bilateral perfusion of half of the volume (infusion of 8 microliters)of the STN with muscimol (8.8 mM) and gadolinium-DTPA ([1 mM] in off and on medication states on sequential days). The second cohort will undergo bilateral perfusion of the entire of the volume (infusion of 16 microliters) of the STN with muscimol (8.8 mM) and gadolinium-DTPA ([1 mM] in off and on medication states on sequential days). Distribution of muscimol using a surrogate imaging tracer (gadolinium-DPTA) will be tracked using real-time MR-imaging and correlated to clinical effect. After the infusions are completed, the catheters will be removed and patients will undergo placement of bilateral STN DBS. Patients will be evaluated using standard PD rating scales to determine the effects to STN neuronal suppression and to compare the effects of muscimol pharmacologic neuronal suppression to DBS effects.

Outcome measures: To determine the distribution of muscimol in the STN and to provide an anatomic correlate for clinical effects of neuronal suppression, real-time 3D-volumetric MR-imaging will be used during infusions. To assess safety, tolerability and clinical effects of muscimol infusion, standard PD rating scales (motor subsection of the Unified PD Rating Scale, timed-up-and-go gait assessment and peg board bradykinesia testing) will be performed following infusion and correlated to real-time infusion MR-imaging studies. To compare the effects of muscimol infusion to STN DBS, the assessments obtained during infusion will be compared to the similar assessment 6 months after DBS placement.

ELIGIBILITY:
* INCLUSION CRITERIA:

Diagnosed with idiopathic PD by UK criteria:

Bradykinesia: At least one of the following:

1. Muscular rigidity
2. 4-6 Hz resting tremor
3. Postural instability not caused by primary visual, vestibular, cerebellar or proprioceptive dysfunction

Three or more required in addition to above for the diagnosis of idiopathic PD:

1. Unilateral onset
2. Rest tremor present
3. Progressive disorder
4. Persistent asymmetry affecting side of onset most
5. Excellent response (70-100%) to levodopa
6. Severe levodopa-induced chorea
7. Levodopa response for 5 years or more
8. Clinical course of ten years or more

   The above clinical features must not be due to trauma, brain tumor, infection, cerebrovascular disease, other known neurological disease (e.g., multiple system atrophy, progressive supranuclear palsy, striatonigral degeneration, Huntington s disease, Wilson s disease, hydrocephalus) or due to known drugs, chemicals or toxicants.

   Disability present despite optimal antiparkinsonian medication therapy.

   Unequivocal responsiveness to levodopa, based on the single-dose levodopa test (as described in the CAPIT and CAPSIT guidelines). In addition to a 33% or greater improvement in one of the timed tasks, a 30% or greater improvement in the UPDRS total motor score will be required to establish unequivocal responsiveness to levodopa.

   Patients must demonstrate at least 6 hours of non-on time and medication side-effects such as levodopa-induced dyskinesias or motor fluctuations.

   Neuropsychological evaluation does not indicate substantial depression or cognitive dysfunction.

   Able to provide proper Informed Consent.

   EXCLUSION CRITERIA:

   Presence of prominent oculomotor palsy, cerebellar signs, vocal cord paresis, orthostatic hypotension (> 20 mm Hg drop on standing), pyramidal tract signs or amyotrophy.

   Presence of dementia (Clinical Dementia Rating Scale score > 1.0 or Mini Mental Status Examination Score < 25).

   Presence or history of psychosis, including if induced by anti-PD medications.

   Presence of untreated or suboptimally treated depression (Hamilton Depression Scale score >10) or a history of a serious mood disorder (for example, requiring psychiatric hospitalization or a prior suicide attempt).

   Presence of substance (drug, alcohol) abuse.

   Presence of hypointensity in the striatum on T2-weighted MR-imaging.

   Contraindication to MR-imaging and/or gadolinium.

   Coagulopathy, anticoagulant therapy, low platelet count, or inability to temporarily stop any antithrombotic medication.

   Prior brain surgery, including gene therapy, radiofrequency ablation or deep brain stimulation.

   Male or female with reproductive capacity who is unwilling to use contraception throughout the study.

   History of stroke or poorly controlled cardiovascular disease.

   Uncontrolled hypertension or diabetes or any other acute or chronic medical condition that would increase the risks of a neurosurgical procedure.

   Clinically active infection, including acute or chronic scalp infection.

   Received investigational agent within 12 weeks prior to screening.

   Unable to comply with the procedures of the protocol, including frequent and prolonged follow-up.

   Baseline hematology, chemistry or coagulation values out of normal range unless not clinically significant with respect to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06-02; Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Determine potential effectiveness of PD symptom reversal by muscimol infusion. Effectiveness will be determined by improvements in (off) and (on) scale UPDRS scores (motor subsection), pegboard testing of bradykinesia and TGUG gait assessment.

SECONDARY OUTCOMES:
Determine feasibilty of distributing muscimol by CED in the STN of PD patients. This endpoint will be the MR-imaging confirmation of distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Kareem A Zaghloul, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)

REFERENCES:
- [Background] Baraldi M, Grandison L, Guidotti A. Distribution and metabolism of muscimol in the brain and other tissues of the rat. Neuropharmacology. 1979 Jan;18(1):57-62. doi: 10.1016/0028-3908(79)90009-1. No abstract available. PMID 418955
- [Background] Bergman H, Wichmann T, DeLong MR. Reversal of experimental parkinsonism by lesions of the subthalamic nucleus. Science. 1990 Sep 21;249(4975):1436-8. doi: 10.1126/science.2402638.
- [Background] Bergman H, Wichmann T, Karmon B, DeLong MR. The primate subthalamic nucleus. II. Neuronal activity in the MPTP model of parkinsonism. J Neurophysiol. 1994 Aug;72(2):507-20. doi: 10.1152/jn.1994.72.2.507. PMID 7983515